CLINICAL TRIAL: NCT00480376
Title: Ofloxacin vs. Gentamicin as Prophylaxis Prior Transrectal Biopsy of Prostate
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 230105
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Infection
Keywords: transrectal biopsy; prostate; prophylaxis antibiotic
MeSH Terms: conditions — Infections | interventions — Ofloxacin; Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ofloxacin
Drug: gentamicin

SUMMARY:
Prostate biopsy is usually conducted transrectal, ultrasonography guided. Since the area is not sterile, infection can be induced during the procedure.

Prophylaxis antibiotic against gram-negative bacteria decreased significantly the amount of infections. Quinolones are considered preferred treatment but there is already an increase in resistance rates. TMP-SMX can not be used empirically due to a high percent of resistant uropathogens. One of the options is aminoglycosides, especially gentamicin. Advantages: very low resistance rate in the community, high concentration is urinary tract, slow clearance, no resistance developed under treatment, chip and with very few side effects.

DETAILED DESCRIPTION:
Prostate biopsy is usually conducted as an ambulatory transrectal needle aspiration, ultrasonography guided. The area is not sterile, with high concentration of gram-negative and anaerobic pathogens, infection can be induced during the procedure to the urinary tract, and even cause bacteremia.

Prior studies concluded that prophylaxis antibiotic against gram-negative bacteria decreased significantly the amount of infections and hence it is accepted to give prophylaxis antibiotics which will cover especially gram-negative bacteria. Other studies show decrease in infections percent in patients that received prophylaxis opposed to those who did not, from 5-30% to less than 1%. Yet, there was no significant difference between those who received one dose and those who were treated for 3-5 days. Quinolones are considered preferred treatment since they can be given orally, but there is already an increase in resistance rates. TMP-SMX can not be used empirically due to a high percent of resistant uropathogens. One of the options is aminoglycosides, especially gentamicin. Advantages: very low resistance rate in the community, high concentration is urinary tract, slow clearance, no resistance developed under treatment, chip and with very few side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients going under transrectal biopsy of prostate with sterile urine culture.

Exclusion Criteria:

* Urine culture not sterile

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2007-06; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
no infection | 48 hours

SECONDARY OUTCOMES:
no infection | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Genady Zelychenko, MD, Principal Investigator — Ha'Emek Medical Center, Afula, Israel
Locations (1):
- Urology outpatient clinic, HaEmek MC, Afula, Israel